CLINICAL TRIAL: NCT07039474
Title: The Application of 18F-G1 PET/CT Targeting Granzyme B in the Pan-cancer Immunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025R0069
Record Dates: First submitted 2025-05-26; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors and Hematological Tumors
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: 18F-G1 — 18F-G1 is injected intravenously with a dose of 0.06-0.08mCi/kg

SUMMARY:
The purpose of this study is to explore the effectiveness of 18F-G1 PET/CT in patients with solid tumors and hematological malignancies receiving immunotherapy

DETAILED DESCRIPTION:
It is urgent to select patients who will benefit from immunotherapy, so as to help the clinicians adjust the regimens and avoid unnecessary side effect. 18F-G1 is a new radioactive tracer targeting granzyme B, holding great promise in assessing early response to immunotherapy. This study will explore the safety of 18F-G1 PET/CT in patients with solid tumors and hematological tumors receiving immunotherapy, analyze its imaging features, and assess its efficacy in predicting early immunotherapy response and prognosis, so as to aid the clinicians in precise patient stratification and regimen adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with a malignant tumor by histopathology who are going to receive immunotherapy (monotherapy or combined immunotherapy) recommended by the multidisciplinary team.
2. Subjects didn't receive previous immunotherapy.
3. There exists at least one measurable target lesion according to the RECIST 1.1.
4. ECOG performance status≤2.
5. The expected survival time is ≥6 months.
6. Effective contraceptive measures will be adopted during the study period and within 6 months after the study.
7. Willing and able to fully understand and sign the informed consent form.

Exclusion Criteria:

1. Women in the preconception period, pregnancy, or lactation period.
2. Combined with other malignant tumor.
3. Diagnosed with autoimmune disease, or have long history of systemic steroid hormone therapy or immunosuppressive therapy.
4. Having a history of severe cardiovascular disease, severe hepatic and renal insufficiency.
5. Receiving radiotherapy or interventional therapy during the immunotherapy.
6. 18F-G1 PET/CT or 18F-FDG PET/CT is not performed in our department, or the interval between baseline imaging and immunotherapy is more than 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with a malignant tumor (solid tumor or hematological tumor) by histopathology who are going to receive immunotherapy (monotherapy or combined immunotherapy).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 18F-G1-related adverse events (AEs). | 3 days after the injection of 18F-G1
  The absolute number of participants with AEs after the injection of 18F-G1 according to CTCAE 5.0.
The vivo accumulation and distribution of 18F-G1 in tumors and major healthy organs. | 40-60 minutes after the injection of 18F-G1
  The accumulation and distribution of 18F-G1 in tumors and major healthy organs, such as liver, lung, kidney, will be quantitatively and qualitatively examined.
the granzyme B specificity of 18F-G1 | 3 years
Assessing the early predictive value of 18F-G1 PET/CT for immunotherapy response. | 6 months
  Participants' overall response will be assessed by RECIST 1.1 criteria or Lugano criteria at the time point of 6 months after immunotherapy. The tumor uptake of 18F-G1 will be compared between the responders and non-responders.

SECONDARY OUTCOMES:
Evaluate the correlation of 18F-G1 accumulation in tumors to long term survival after immunotherapy. | 3 years
  Participants will be categorized into groups with high or low 18F-G1 uptake in tumor lesions. The progression-free survival (PFS) as assessed by RECIST 1.1 criteria or Lugano criteria will be compared between the two groups.

IPD SHARING:
Plan to Share IPD: No